CLINICAL TRIAL: NCT06859229
Title: Effects on Gait Patterns of a New Technological Pathway for Gait Rehabilitation in Patients with Movement Disorders
Brief Title: New Technological Pathway for Gait Rehabilitation
Acronym: LABODIMOTO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 45/2020
Record Dates: First submitted 2025-01-23; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Neurological Diseases or Conditions; Cardiovascular Diseases; Neuromuscular Disease
Keywords: neurorehabilitation; gait rehabilitation; analysis of movement; neuroplasticity
MeSH Terms: conditions — Cardiovascular Diseases; Neuromuscular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Innovative gait rehabilitation pathway (Experimental): The group will be treated with a dynamic pathway with advanced technology for gait rehabilitation.
  Interventions: Device: Innovative technology pathway for gait neurorehabilitation
- Conventional gait rehabilitation (Active Comparator): The group will be treated with conventional gait rehabilitation strategies.
  Interventions: Other: Conventional gait rehabilitation strategy

INTERVENTIONS:
Device: Innovative technology pathway for gait neurorehabilitation — Participants will be assigned to either an advanced or traditional training pathway based on the protocol. The innovative tehcnology pathway for gait rehabilitation will incorporate devices such as exoskeletons, virtual reality systems, and body-weight suspension (BWS) devices to enhance gait rehabilitation. At the end of the training period, participants will undergo follow-up evaluation tests to assess outcomes.
  Other Names: Robotic rehabilitation; virtual reality rehabilitation
  Arms: Innovative gait rehabilitation pathway
Other: Conventional gait rehabilitation strategy — The control group will undergo a traditional rehabilitation program that follows standard clinical protocols for gait recovery. This program will include conventional therapeutic exercises aimed at improving strength, balance, coordination, and functional mobility
  Other Names: Gait rehabilitation; conventional neurorehabilitation
  Arms: Conventional gait rehabilitation

SUMMARY:
**Brief Summary**

The study aims to explore how the integration of visual and motor systems can be trained and enhanced to improve gait rehabilitation in patients with various neurological and cardiovascular conditions. Scientific evidence highlights that physical activity requires coordination and precise processing of visual, auditory, and sensory information from the external environment, which is then integrated at the brain level. This process establishes synaptic connections that direct the movement of arms, hands, legs, and the trunk through bottom-up and top-down mechanisms. However, inaccurate or incomplete perceptual information can impair performance, even when accurate visual stimuli are provided, emphasizing the importance of assessing and enhancing visuo-motor integration.

The research investigates the central mechanisms controlling peripheral muscle activation patterns during gait. While over-ground walking in healthy individuals generally does not activate the prefrontal cortex except in dual-task scenarios, evidence suggests that post-stroke patients exhibit increased prefrontal cortex metabolism during walking. Recent studies have shown that gait training with exoskeletal systems improves walking patterns in post-stroke patients by altering muscle activation patterns and increasing fronto-parietal connectivity.

This study seeks to answer the following question: How do central and peripheral mechanisms interact to influence gait rehabilitation outcomes, and what role do visuo-motor integration and neuroplasticity play in this process? To address this, advanced neuroimaging technologies such as fMRI, dtMRI, and NIRS will be employed to investigate these mechanisms in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a Montreal Cognitive Assessment (MoCA) score, corrected for age and education, equal to or greater than 20.
* Subjects capable of walking independently (Functional Ambulation Categories - FAC > 2).

Exclusion Criteria:

* Cognitive impairments that compromise the understanding and/or execution of the proposed exercises.
* Associated comorbidities that prevent maintaining an upright position or walking (e.g., hypotension).
* Refusal or inability to provide informed consent.
* Patients with contraindications to the use of the technological equipment required for the dynamic movement pathway.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Neural correlates of movement | From enrollment to end of treatment at five weeks
  We will assess motor functions using clinical scales (e.g., Fugl-Meyer Lower Extremity), to explore potential links between gait rehabilitation and motor recovery.
  Time Frame: Baseline (T0), post-intervention (T1, 12 weeks after baseline), and follow-up (T2, 3 months post-intervention).

SECONDARY OUTCOMES:
Neurophysiological outcome | From enrollment to end of treatment at five weeks
  A secondary objective is to investigate the neurophysiological changes associated with the intervention. This includes analyzing EEG parameters (such as changes in alpha, theta, and beta rhythms) to understand the underlying mechanisms driving motor improvements.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro Neurolesi Bonino-Pulejo, Messina, Maine, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hidler J, Nichols D, Pelliccio M, Brady K, Campbell DD, Kahn JH, Hornby TG. Multicenter randomized clinical trial evaluating the effectiveness of the Lokomat in subacute stroke. Neurorehabil Neural Repair. 2009 Jan;23(1):5-13. doi: 10.1177/1545968308326632. PMID 19109447
- [Background] Hornby TG, Campbell DD, Kahn JH, Demott T, Moore JL, Roth HR. Enhanced gait-related improvements after therapist- versus robotic-assisted locomotor training in subjects with chronic stroke: a randomized controlled study. Stroke. 2008 Jun;39(6):1786-92. doi: 10.1161/STROKEAHA.107.504779. Epub 2008 May 8. PMID 18467648
- [Background] Chang WH, Kim YH. Robot-assisted Therapy in Stroke Rehabilitation. J Stroke. 2013 Sep;15(3):174-81. doi: 10.5853/jos.2013.15.3.174. Epub 2013 Sep 27. PMID 24396811